CLINICAL TRIAL: NCT00028600
Title: Autologous Followed By Non-Myeloablative Allogeneic Transplant For Multiple Myeloma
Brief Title: Peripheral Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-100001; U10CA031946 (NIH); CALGB-100001; CDR0000069109 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; betibeglogene autotemcel; Cyclophosphamide; fludarabine phosphate; Melphalan; Methotrexate; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous + Allogeneic Transplant (Experimental): autologous PB stem cell transplant followed by non-myeloablative allogeneic transplant fr multiple myeloma
  Interventions: Biological: filgrastim; Biological: CD34+ cells; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: melphalan; Drug: methotrexate; Drug: tacrolimus

INTERVENTIONS:
Biological: filgrastim — PBSC collection: 10 ug/kg/d subQ inj D 5 until completion of collection Auto transpl: 5 ug/kg/d subQ inj D 5 until ANC >= 1500/uL for 2d or 5000/uL for 1 d Allo transpl: 5ug/kg/d subQ inj D 7 until ANC > 1000/uL for 3 days Donor pheresis: 10ug/kg/d subQ inj d -5 thru -2
  Other Names: G-CSF
Biological: CD34+ cells — 2-8,000,000/kg IV infusion allogeneic transplant 2,000,000/kg IV infusion autologous transplant
Drug: cyclophosphamide — 4g/sq m IV infusion over 1-2 hrs D 1 for auto, and 1g/sq m/d IV infusion over 1 hr on D -4 thru -3 for allo, transplant prep
Drug: fludarabine phosphate — 30mg/sq m/d IVPB over 30 min d -7 thru -3 allo transpl
Drug: melphalan — 200mg/sq m IV infusion over 15-30 min D 2 auto transpl
Drug: methotrexate — 5mg/sq m/d IV infusion D 1,3,& 6: allo transpl
Drug: tacrolimus — 0.03mg/kg PO bid starting dose, D -1 thru +90, then taper thru D +150

SUMMARY:
RATIONALE: Peripheral blood stem cell transplant using stem cells from the patient or a donor may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells. The donated stem cells may also help destroy any remaining cancer cells (graft-versus-tumor effect).

PURPOSE: This phase II trial is studying how well autologous peripheral stem cell transplant followed by donor peripheral stem cell transplant works in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether autologous peripheral blood stem cell transplantation (PBSCT) followed by non-myeloablative allogeneic PBSCT is associated with no more than 20% treatment-related mortality rates at 6 months in patients with multiple myeloma.
* Determine the response rate of patients treated with this regimen.
* Determine the percent donor chimerism in patients treated with this regimen.
* Determine the rate of graft-vs-host disease in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the disease-free and overall survival of patients treated with this regimen.
* Determine whether abnormal cytogenetics at presentation correlate with poor response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive cyclophosphamide IV over 1-2 hours on day 1 and filgrastim (G-CSF) subcutaneously (SC) beginning on day 5 and continuing until peripheral blood stem cell (PBSC) collection is complete.

Approximately 2-4 weeks after PBSC collection, patients receive melphalan IV over 15-30 minutes on day -2. Patients then undergo autologous PBSC transplantation (PBSCT) on day 0. Patients receive G-CSF SC beginning on day 5 and continuing until blood counts recover.

Approximately 2-4 months after autologous PBSCT, patients receive fludarabine IV over 30 minutes on days -7 to -3 and cyclophosphamide IV over 1 hour on days -4 to -3. Patients undergo allogeneic PBSCT on day 0. Patients receive G-CSF SC beginning on day 7 and continuing until blood counts recover.

Patients receive graft-vs-host disease (GVHD) prophylaxis comprising oral tacrolimus twice daily on days -1 to 90 followed by a taper on days 91-150 and methotrexate IV on days 1, 3, and 6.

After day 120, patients with stable or progressive disease and no evidence of active GVHD may receive donor lymphocyte infusion (DLI) over 2 hours. Patients may receive up to 3 DLIs every 8 weeks.

Patients are followed every 3 months for 3 years, every 6 months for 5 years, and then annually for 15 years.

PROJECTED ACCRUAL: A maximum of 63 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of active multiple myeloma that requires treatment

  * Durie-Salmon stage I, II, and III
* No more than 1 progression after initial therapy
* Must have HLA-identical sibling donor (6/6) by serologic typing (A, B, DR)

  * No syngeneic donors
* Must also be enrolled on protocol CLB-8461 (Cytogenetic Studies in Acute Leukemia)

PATIENT CHARACTERISTICS:

Age:

* Under 65

Performance status:

* NCI CTC 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 500/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin less than 2 mg/dL
* AST less than 3 times upper limit of normal (ULN)
* Alkaline phosphatase less than 3 times ULN

Renal:

* Creatinine less than 2 mg/dL
* Creatinine clearance greater than 40 mL/min

Cardiovascular:

* LVEF at least 30% by MUGA scan

Pulmonary:

* DLCO greater than 40% of predicted
* No symptomatic pulmonary disease

Other:

* HIV negative
* No uncontrolled diabetes mellitus
* No active serious infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* Prior alkylating-agent therapy allowed if no more than 12 months duration

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* At least 4 weeks since prior surgery

Other:

* All prior therapy no more than 18 months duration

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2001-11; Primary Completion 2006-06 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Treatment-related mortality | 6 months

SECONDARY OUTCOMES:
Treatment Completion Rate | post treatment
Respone Rate | 2-4 wks prior, and 3,6 mon then q 3 mon for 3 yrs, post allo transpl, then q 6 mon for max 15 yrs from study entry
Chimerism Rate | 1,2,3,4, & 6 mon post allo transpl, & 100 d post DLI
GVHD Incidence | post allo transpl, & pre & post DLI
Survival | 2 years
  Overall and disease free survival will be assessed
Correlation of cytogenetics and response | 6, 12 mon then q 1 yr for 3 yrs post allo transpl

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C. Anderson, MD, Study Chair — Dana-Farber Cancer Institute
Locations (15):
- United States (15):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - Saint Louis, St Louis, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Holstein SA, Suman VJ, Owzar K, Santo K, Benson DM Jr, Shea TC, Martin T, Silverman M, Isola L, Vij R, Cheson BD, Linker C, Anderson KC, Richardson PG, McCarthy PL. Long-Term Follow-up of CALGB (Alliance) 100001: Autologous Followed by Nonmyeloablative Allogeneic Transplant for Multiple Myeloma. Biol Blood Marrow Transplant. 2020 Aug;26(8):1414-1424. doi: 10.1016/j.bbmt.2020.03.028. Epub 2020 Apr 20. PMID 32325171